CLINICAL TRIAL: NCT07396116
Title: Preoperative Hypofractionated Radiotherapy Combined With Immunotherapy Followed by Surgery for Retroperitoneal Sarcoma (FUSION-02)
Brief Title: Preoperative Hypofractionated RT + Immunotherapy & Surgery for Retroperitoneal Sarcoma (FUSION-02)
Acronym: FUSION-02
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, NINGNING LU, Principle Investigator, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC FUSION-02
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Soft Tissue Sarcoma (STS); Retroperitoneal Sarcoma; Immunotherapy; Radiotherapy Side Effect; Ultra-hypofractionated Radiotherapy
Keywords: hypofractionated radiotherapy; retroperitoneal sarcoma; soft tissue sarcoma; immunotherapy; peri-operative complications
MeSH Terms: conditions — Sarcoma; Radiation Injuries | interventions — Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypofractionated Radiotherapy Combined with Immunotherapy (Experimental): Patients receive hypofractionated radiotherapy with 43.5Gy in 15 fractions, combined with immunotherapy, followed by surgery done at 6-10 weeks post-radiotherapy (RT).
  Interventions: Radiation: ultra-hypofractionated radiotherapy combined with immunotherapy

INTERVENTIONS:
Radiation: ultra-hypofractionated radiotherapy combined with immunotherapy — ultra-hypo-fractionated radiotherapy with 43.5Gy in 15 fractions combined with immunotherapy, followed by surgery done at 6 to 10 weeks post-RT

SUMMARY:
To investigate the feasibility and peri-operative complications of preoperative hypo-fractionated radiotherapy combined with immunotherapy followed by surgery for retroperitoneal sarcoma

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis & Indication: Primary or recurrent abdominopelvic soft tissue sarcoma. Patients are deemed to have a high probability of R1/R2 resection with upfront surgery and are confirmed to require radiotherapy following Multidisciplinary Team (MDT) discussion.
* Target Volume: In cases of multifocal disease, all lesions must be safely encompassable within a single radiotherapy target volume.
* Age: Age ≥ 18 years.
* Performance Status: Eastern Cooperative Oncology Group (ECOG) performance status 0-2; American Society of Anesthesiologists (ASA) score ≤ 2; patients must be expected to tolerate surgery and radiotherapy.
* Pathology: Histologically confirmed soft tissue sarcoma.
* Measurability: Presence of evaluable lesions.
* Life Expectancy: Life expectancy > 5 years.
* Hematological & Hepatic Function: Adequate organ function
* Renal Function: Adequate renal function defined as Glomerular Filtration Rate (GFR) ≥ 50 ml/min (calculated by Cockcroft-Gault formula), and split renal function imaging confirms function in the contralateral kidney.
* Contraception: Female patients of childbearing potential, or male patients with female partners of childbearing potential, must agree to use effective contraception during the entire treatment period and for 6 months after the last dose.
* Consent: Signed informed consent form.
* Follow-up: Capable of complying with follow-up requirements.

Exclusion Criteria:

* Significant Comorbidities: Patients with the following concurrent conditions: active hemorrhage, ulceration, intestinal perforation, intestinal obstruction, uncontrolled hypertension, cardiac insufficiency (NYHA Class III-IV), severe hepatic or renal dysfunction (Grade 4), mesenteric ischemia, or severe inflammatory bowel disease (IBD).
* Excluded Histologies: Other pathological types, including Gastrointestinal Stromal Tumor (GIST), sarcomatoid carcinoma, sarcomas primarily treated with chemotherapy (e.g., rhabdomyosarcoma and PNET), desmoid fibromatosis, and benign tumors.
* Unresectability: Tumor invasion into critical structures such as the liver, pancreatic head, or abdominal aorta, rendering the tumor deemed unresectable.
* Prior Radiotherapy: History of prior radiotherapy to the same anatomical region.
* Distant Metastasis: Presence of distant metastasis (M1) confirmed by comprehensive imaging/examination within 4 weeks prior to enrollment.
* Contraindications to Surgery/Protocol: Presence of other severe medical comorbidities that contraindicate surgery or preclude participation in the study.
* Planned Neoadjuvant Chemotherapy: Patients scheduled to receive (concurrent) neoadjuvant chemotherapy.
* Recent Systemic Therapy: Receipt of chemotherapy or other systemic treatments within 4 weeks prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-02-12 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Peri-operative complications | From surgery date up to 7 days later
  The proportion of patients who suffer from

CONTACTS AND LOCATIONS:
Locations (1):
- Radiotherapy Department of Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided